CLINICAL TRIAL: NCT04659915
Title: Counteracting Deleterious Metabolic Glucocorticoid Effects With Metformin - A Double-blind, Randomized, Placebo-controlled, Cross-over Study
Brief Title: Counteracting Deleterious Metabolic Glucocorticoid Effects With Metformin
Acronym: Gluco-Met
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eleonora Seelig (Other)
Responsible Party: Sponsor-Investigator, Eleonora Seelig, Principal Investigator, University Hospital, Basel, Switzerland
Organization: University Hospital, Basel, Switzerland (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: EKNZ 2020-01233
Record Dates: First submitted 2020-12-01; First posted 2020-12-09 (Actual); Last update posted 2021-09-23 (Actual); Status verified 2021-09

CONDITIONS: Glucocorticoid Effect
MeSH Terms: interventions — Metformin; Prednisone

STUDY DESIGN:
Intervention Model Description: Double-blind, randomized, placebo-controlled cross-over study
Who Masked: Participant, Investigator
Masking Description: Placebo-controlled
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Metformin + Prednison (Experimental): During one of the study periods, subjects receive Metformin 500 mg tablets p.o. for seven days (starting with a dose of 500 mg /d, then the dose will be increased by 500 mg the next days until 2000 mg /d is achieved).
  Subjects also receive Prednisone 20 mg 1.5x/d tablets p.o. for seven days.
  Interventions: Drug: Metformin 500 mg Oral Tablets + Prednisone 20mg Tablets
- Placebo + Prednison (Placebo Comparator): During the other study period, subjects receive the same dose of placebo tablets p.o instead of metformin. Subjects also receive Prednisone 20 mg 1.5x/d tablets p.o. for seven days.
  Interventions: Drug: Placebo 500 mg Tablets + Prednisone 20mg Tablets

INTERVENTIONS:
Drug: Metformin 500 mg Oral Tablets + Prednisone 20mg Tablets — During one phase of the study: Metformin 500mg Day 1 1-0-0 Day 2 1-0-0 Day 3 1-0-1 Day 4 1-0-1 Day 5 2-0-1 Day 6 2-0-1 Day 7 4-0-0
  In combination with prednisone 20mg: day 1 to day 7 1.5-0-0.
  Arms: Metformin + Prednison
Drug: Placebo 500 mg Tablets + Prednisone 20mg Tablets — During another phase of the study: identical looking placebo pills starting day 1 500mg 1-0-0, day 2 500mg 1-0-0, day 3 500mg 1-0-1, day 4 500mg 1-0-1, day 5 500mg 2-0-1. day 6 2-0-1, day 7 4-0-0. In combination with prednisone 20mg: day 1 to day 7 1.5-0-0.
  Arms: Placebo + Prednison

SUMMARY:
Supraphysiological doses of glucocorticoids (GCs) are widely prescribed as immunosuppressants and metabolic side effects such as obesity and diabetes are extremely common. Efforts to investigate and prevent these side effects are lacking. The antidiabetic drug metformin was shown in previous studies to prevent deterioration of glucose homeostasis during GC therapy in patients. However, mechanisms of metformin counteracting GC-induced side effects remain poorly understood.

In a randomized, placebo-controlled, cross-over study, 18 healthy volunteers will receive a 7-day course of prednisone with metformin or placebo. Established methods will be used to assess systemic changes in energy homeostasis and novel techniques such as metabolomics will identify underlying pathways. This will advance the understanding of energy homeostasis during GC excess, may prevent thousands of patients from GC-induced side effects and also offers a model for targeting disrupted endogenous GCs secretion.

DETAILED DESCRIPTION:
Obesity is one of the most serious health problems in the 21st century (1). Currently, more than 700 million people world-wide are obese and face an increased risk of morbidity and a reduced life-expectancy of up to 10 years (1, 2). High energy food and a sedentary lifestyle are driving the current obesity pandemic (3). Sleep deprivation and psychological stress also have been identified as contributing factors (4). Many of these factors activate the hypothalamic-pituitary-adrenal (HPA) axis, the key regulatory pathway of energy homeostasis. Activation of the HPA-axis leads to secretion of glucocorticoids (GCs) from the adrenal glands. GCs control energy homeostasis by mobilizing and redistributing energy substrates (5). In an evolutionary context, GCs are particularly important during periods of stress, especially when food is scarce. In today's environment, where food is abundantly available, GCs potentially can become deleterious by severely disrupting energy homeostasis. Therefore, the GC pathway has gained interest as a potential treatment target for the metabolic syndrome.

Next to their essential role in energy homeostasis, glucocorticoids are the most commonly prescribed immunosuppressant drugs. GCs are used for acute as well as chronic conditions in virtually all medical disciplines (6). It is well known that patients on GC treatment are at high risk for developing numerous side effects. Next to dyslipidaemia, arterial hypertension and cardiovascular disease, up to 80% of patients experience weight gain, while around 40% develop diabetes (7). Currently, no therapies exist to prevent any of these side effects. The only available strategy to prevent GC-induced side effects is to restrain GC use.

The objective of this project is to test in a clinical study in humans whether metformin can counteract the deleterious metabolic effects developed after a short-term glucocorticoid treatment. The primary objective is to test how metformin counteracts metabolic side effects of GCs compared to placebo. Secondary objectives are to detect underlying pathways in blood (metabolomics), adipose tissue (gene expression analysis) and mitochondria (Cytosensor) with metformin in combination with prednisone compared to placebo and prednisone.

This is a double-blind, randomized, placebo-controlled cross-over study. After screening, subjects will be randomized to two crossover 7-day study periods with a washout period of 28 days:

A) Participants will receive prednisone 30 mg/d p.o. and metformin (starting with a dose of 500 mg/d and increasing the dose by 500 mg every other day until 2000 mg/d are achieved).

B) Participants will receive prednisone 30 mg/d p.o. and placebo p.o. (starting with a dose of 500 mg/d and increasing the dose by 500 mg every other day until 2000 mg/d are achieved).

ELIGIBILITY:
Inclusion Criteria:

* BMI 18.5 - 25 kg/m2

Exclusion Criteria:

* Any current significant disease,
* Any medication
* Glucocorticoids and/ or metformin for up to four weeks before study inclusion
* Regular alcohol intake (>30g/d),
* Regular physical activity (>4hrs per week),
* Known allergy to metformin,
* Inability or unwillingness to provide informed consent.

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Since hormone fluctuations associated with the menstrual cycle may alter cortisol levels, women will not be included in the study. Although diversity will be reduced and the statements of the study cannot be applied to the female sex, these strict inclusion criteria allow an optimal homogeneity and increase statistical power.
Enrollment: 19 (Actual)
Dates: Start 2021-02-25 (Actual); Primary Completion 2021-08-18 (Actual); Study Completion 2021-08-18 (Actual)

PRIMARY OUTCOMES:
Insulin sensitivity | Two 1-week intervention periods
  Change in insulin sensitivity (HOMA-Index) assessed with a mixed meal tolerance test.

SECONDARY OUTCOMES:
Lipids (mmol/l) | Two 1-week intervention periods
  Blood sample
Cortisol (nmol/l) | Two 1-week intervention periods
  Blood sample
GLP-1 (nmol/l) | Two 1-week intervention periods
  Blood sample
GIP (nmol/l) | Two 1-week intervention periods
  Blood sample
PYY (pg/ml) | Two 1-week intervention periods
  Blood sample
C-peptide (pmol/l) | Two 1-week intervention periods
  Blood sample
T3 (nmol/l) | Two 1-week intervention periods
  Blood sample
T4 (nmol/l) | Two 1-week intervention periods
  Blood sample
TSH (mIU/l) | Two 1-week intervention periods
  Blood sample
HGH (mIU/l) | Two 1-week intervention periods
  Blood sample
Sympathetic nervous system activity | Two 1-week intervention periods
  Heart rate variability analysis
Blood pressure | Two 1-week intervention periods
  Assessment of blood pressure with a standard blood pressure monitor.
Weight | Two 1-week intervention periods
  Measurement of weight with a standard scale
Energy expenditure | Two 1-week intervention periods
  Basal metabolic rate measured with indirect calorimetry
Substrate utilisation | Two 1-week intervention periods
  Respiratory quotient assessed with indirect calorimetry
GDF-15 (pg/mL) | Two 1-week intervention periods
  Blood sample

OTHER OUTCOMES:
Metabolomics | Two 1-week intervention periods
  Metabolomics will be performed in blood plasma
Gene expression analysis | Two 1-week intervention periods
  Adipose tissue biobsy

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Basel, Basel, Canton of Basel-City, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] GBD 2015 Obesity Collaborators; Afshin A, Forouzanfar MH, Reitsma MB, Sur P, Estep K, Lee A, Marczak L, Mokdad AH, Moradi-Lakeh M, Naghavi M, Salama JS, Vos T, Abate KH, Abbafati C, Ahmed MB, Al-Aly Z, Alkerwi A, Al-Raddadi R, Amare AT, Amberbir A, Amegah AK, Amini E, Amrock SM, Anjana RM, Arnlov J, Asayesh H, Banerjee A, Barac A, Baye E, Bennett DA, Beyene AS, Biadgilign S, Biryukov S, Bjertness E, Boneya DJ, Campos-Nonato I, Carrero JJ, Cecilio P, Cercy K, Ciobanu LG, Cornaby L, Damtew SA, Dandona L, Dandona R, Dharmaratne SD, Duncan BB, Eshrati B, Esteghamati A, Feigin VL, Fernandes JC, Furst T, Gebrehiwot TT, Gold A, Gona PN, Goto A, Habtewold TD, Hadush KT, Hafezi-Nejad N, Hay SI, Horino M, Islami F, Kamal R, Kasaeian A, Katikireddi SV, Kengne AP, Kesavachandran CN, Khader YS, Khang YH, Khubchandani J, Kim D, Kim YJ, Kinfu Y, Kosen S, Ku T, Defo BK, Kumar GA, Larson HJ, Leinsalu M, Liang X, Lim SS, Liu P, Lopez AD, Lozano R, Majeed A, Malekzadeh R, Malta DC, Mazidi M, McAlinden C, McGarvey ST, Mengistu DT, Mensah GA, Mensink GBM, Mezgebe HB, Mirrakhimov EM, Mueller UO, Noubiap JJ, Obermeyer CM, Ogbo FA, Owolabi MO, Patton GC, Pourmalek F, Qorbani M, Rafay A, Rai RK, Ranabhat CL, Reinig N, Safiri S, Salomon JA, Sanabria JR, Santos IS, Sartorius B, Sawhney M, Schmidhuber J, Schutte AE, Schmidt MI, Sepanlou SG, Shamsizadeh M, Sheikhbahaei S, Shin MJ, Shiri R, Shiue I, Roba HS, Silva DAS, Silverberg JI, Singh JA, Stranges S, Swaminathan S, Tabares-Seisdedos R, Tadese F, Tedla BA, Tegegne BS, Terkawi AS, Thakur JS, Tonelli M, Topor-Madry R, Tyrovolas S, Ukwaja KN, Uthman OA, Vaezghasemi M, Vasankari T, Vlassov VV, Vollset SE, Weiderpass E, Werdecker A, Wesana J, Westerman R, Yano Y, Yonemoto N, Yonga G, Zaidi Z, Zenebe ZM, Zipkin B, Murray CJL. Health Effects of Overweight and Obesity in 195 Countries over 25 Years. N Engl J Med. 2017 Jul 6;377(1):13-27. doi: 10.1056/NEJMoa1614362. Epub 2017 Jun 12. PMID 28604169
- [Result] Prospective Studies Collaboration; Whitlock G, Lewington S, Sherliker P, Clarke R, Emberson J, Halsey J, Qizilbash N, Collins R, Peto R. Body-mass index and cause-specific mortality in 900 000 adults: collaborative analyses of 57 prospective studies. Lancet. 2009 Mar 28;373(9669):1083-96. doi: 10.1016/S0140-6736(09)60318-4. Epub 2009 Mar 18. PMID 19299006
- [Result] van der Klaauw AA, Farooqi IS. The hunger genes: pathways to obesity. Cell. 2015 Mar 26;161(1):119-132. doi: 10.1016/j.cell.2015.03.008. PMID 25815990
- [Result] Vgontzas AN, Lin HM, Papaliaga M, Calhoun S, Vela-Bueno A, Chrousos GP, Bixler EO. Short sleep duration and obesity: the role of emotional stress and sleep disturbances. Int J Obes (Lond). 2008 May;32(5):801-9. doi: 10.1038/ijo.2008.4. Epub 2008 Feb 5. PMID 18253159
- [Result] de Guia RM, Rose AJ, Herzig S. Glucocorticoid hormones and energy homeostasis. Horm Mol Biol Clin Investig. 2014 Aug;19(2):117-28. doi: 10.1515/hmbci-2014-0021. PMID 25390020
- [Result] Laugesen K, Jorgensen JOL, Sorensen HT, Petersen I. Systemic glucocorticoid use in Denmark: a population-based prevalence study. BMJ Open. 2017 May 29;7(5):e015237. doi: 10.1136/bmjopen-2016-015237. PMID 28554927
- [Result] McDonough AK, Curtis JR, Saag KG. The epidemiology of glucocorticoid-associated adverse events. Curr Opin Rheumatol. 2008 Mar;20(2):131-7. doi: 10.1097/BOR.0b013e3282f51031. PMID 18349741